CLINICAL TRIAL: NCT06674473
Title: Effect and Evaluation of Long-term Isokinetic Training of Knee Joint Under the Influence of Stiffness
Brief Title: Evaluation of Long-term Isokinetic Training of Knee Joint
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beihang University (Other)
Responsible Party: Principal Investigator, Yuan Fuzhen, Principle Investigator, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-492-04
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Knee Injuries and Disorders
MeSH Terms: conditions — Knee Injuries; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted Rehabilitation (Experimental): In this clinical trial, 6 patients who meet the inclusion criteria will be enrolled in the experimental group to undergo rehabilitation using a portable isokinetic device.
  Interventions: Device: With robot assistance
- None-robot-assisted Rehabilitation (Active Comparator): The control group will consist of 6 patients who meet the inclusion criteria and will undergo traditional bodyweight rehabilitation
  Interventions: Behavioral: traditional bodyweight rehabilitation

INTERVENTIONS:
Device: With robot assistance — Use a portable isokinetic device
  Arms: Robot-assisted Rehabilitation
Behavioral: traditional bodyweight rehabilitation — Use traditional bodyweight rehabilitation
  Arms: None-robot-assisted Rehabilitation

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of isokinetic rehabilitation training under optimal stiffness in patients undergoing knee joint rehabilitation. The main questions it aims to answer are:

* Does isokinetic training under optimal stiffness lead to greater force exertion compared to traditional bodyweight training?
* What are the long-term (6-week) effects of isokinetic training under optimal stiffness on joint flexibility and muscle strength? Researchers will compare the effects of isokinetic training under optimal stiffness to traditional bodyweight training to see if isokinetic training produces superior improvements in muscle strength, flexibility, and overall functional recovery.

Participants will:

* Perform regular training sessions using a portable knee joint isokinetic trainer, customized to their optimal stiffness for maximum force exertion.
* Engage in a 6-week rehabilitation program, with assessments at the beginning, and end of the study to evaluate changes in muscle strength, and functional recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-60 years.
2. Patients with unilateral anterior cruciate ligament (ACL) rupture, with or without meniscus injury.
3. Postoperative period of 3-6 months.
4. No restriction in knee extension or flexion movements.

Exclusion Criteria:

1. Patients with major diseases or conditions such as coronary heart disease, myocardial infarction, heart failure, cerebral infarction, cerebral hemorrhage, or malignant tumors.
2. Pregnant or breastfeeding women and other special populations.
3. Patients who refuse to sign the informed consent form or are unable to complete the entire study process.
4. Patients currently infected with human immunodeficiency virus (HIV), or with a history of infectious hepatitis B or C.
5. Patients with concurrent medical issues, including but not limited to: (1) Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥95 mmHg), congestive heart failure (New York Heart Association functional classification of stage III or IV). (2) Patients with mental incapacity or an inability to comprehend the study requirements.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional area of the quadriceps | Before 1st practice, and after 12th practice (6 weeks * 2 practices/week = 12 practices)
  Using MRI，Up to 6 weeks
Cross-sectional area of the hamstrings | Before 1st practice, and after 12th practice (6 weeks * 2 practices/week = 12 practices)
  using MRI， Up to 6 weeks
Peak flexion and extension knee torque | During each practice (6 weeks * 2 practices/week = 12 practices).
  Using an integrated torque sensor
Average flexion and extension knee torque | During each practice (6 weeks * 2 practices/week = 12 practices).
Flexion and extension knee work | In each ptractice (6 weeks * 2 practices /week = 12 practices).
  Work=Torque*Speed

SECONDARY OUTCOMES:
Thigh circumference | In each ptractice (6 weeks * 2 practices /week = 12 practices).
  10 cm proximal to the superior pole of the patella
Knee joint pain score (VAS score) | Before 1st practice, and after 12th practice (6 weeks * 2 practices/week = 12 practices)
  Up to 6 weeks，max. =100, min. =0, Visual Analogue Scale=VSA, A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT06674473/Prot_SAP_ICF_000.pdf